CLINICAL TRIAL: NCT05711121
Title: Caudal Versus S1 Transforaminal Epidural Steroid Injection for the Treatment of Unilateral S1 Radiculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Collaborators: Marmara University (Other)
Responsible Party: Principal Investigator, Bilinç Doğruöz Karatekin, Bilinc Dugruoz Karatekin, M.D., Department of Physical Medicine and Rehabilitation, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09.2020.719
Record Dates: First submitted 2023-01-09; First posted 2023-02-02 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Lumbosacral Radiculopathy
Keywords: epidural injection; radicular pain; disc herniation; lumbosacral radiculopathy; transforaminal injection; caudal injection
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Intervention Model Description: Patients having radicular pain were randomized to either caudal or transforaminal epidural injection group
Who Masked: Participant, Investigator
Masking Description: Patients and the investigator assessing the treatment results were blinded to the injection technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S1 transforaminal (Active Comparator): The group receiving S1 transforaminal epidural steroid injection
  Interventions: Procedure: Transforaminal epidural steroid injection
- Caudal (Active Comparator): The group receiving caudal epidural steroid injection
  Interventions: Procedure: Caudal epidural steroid injection

INTERVENTIONS:
Procedure: Transforaminal epidural steroid injection — Fluoroscopy-guided transforaminal epidural injection for radicular pain resulting from a disc herniation.
  Arms: S1 transforaminal
Procedure: Caudal epidural steroid injection — Fluoroscopy-guided caudal epidural injection for radicular pain resulting from a disc herniation.
  Arms: Caudal

SUMMARY:
To compare the efficacies of two different interventional techniques (Caudal epidural steroid injection and S1 transforaminal epidural steroid injection) for the treatment of unilateral S1 radiculopathy.

DETAILED DESCRIPTION:
Epidural steroid injections are commonly performed for the treatment of radicular pain resulting from a disc herniation. There are 3 different methods to deliver steroids to epidural area which are caudal, interlaminar and transforaminal routes. Lower lumbar and sacral radiculopathies can be managed with caudal epidural steroid injection which is generally quite easier to perform in comparison to transforaminal injection. Transforaminal epidural injection provides injectate to reach anterior epidural area and is the most target specific technique among others. In the present study investigators aim is to compare the success rates of these two different procedures regarding unilateral S1 radiculopathy. The patients referring to the pain medicine outpatient clinic of a university hospital for unilateral radicular pain and diagnosed S1 radiculopathy were planned to be randomized into these two different intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral radicular pain resulting from a paracentral L5-S1 disc herniation causing S1 nerve root compression.

Exclusion Criteria:

* History of previous surgery, pregnancy, neurological disorders, bleeding diathesis, contrast medium allergy, spinal disorders, rheumatologic diseases

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
50 percent pain relief | 3 months
  Number of patients having at least 50 percent pain relief

SECONDARY OUTCOMES:
Oswestry Disability Index | 3 months
  Improvement in disability scores, 0 is the best, 100 is the worst score.
Procedure time | during procedure
  The overall ease of application regarding procedure time.
Radiation exposure | during procedure
  The exposed radiation dose during the procedures

CONTACTS AND LOCATIONS:
Overall Officials: Osman Hakan Gunduz, Prof., Study Director — Marmara University
Locations (1):
- Marmara University School of Medicine, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Patient data, statistics and study protocol can be shared.
Supporting Information: Study Protocol, SAP
Time Frame: 1 week